CLINICAL TRIAL: NCT01181661
Title: Internet-based Group Contingency Management to Promote Smoking Abstinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jesse Dallery, Principal Investigator, National Development and Research Institutes, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21DA029162 (NIH); 1R21DA029162 (NIH)
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Cigarette Smoking
Keywords: Cigarette; Smoking; Nicotine; Contingency Management; Voucher Reinforcement; Smoking Abstinence; Internet; Internet-based Treatment; Group Contingencies
MeSH Terms: conditions — Cigarette Smoking; Smoking

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full Group Contingency (Experimental): This group (n = 20) will earn vouchers based only on team (n = 4) performance. Only if all members of the team submit a negative sample (CO ≤ 4 ppm), will they each earn a voucher.
  Interventions: Behavioral: Full Group Contingency
- Mixed Group Contingency (Experimental): This group (n = 20) will earn vouchers based on both individual and team (n = 4) performance. If an individual submits a negative sample (CO ≤ 4 ppm), s/he will earn a voucher. Additionally, bonus vouchers will be earned if all team members submit negative samples.
  Interventions: Behavioral: Mixed Group Contingency

INTERVENTIONS:
Behavioral: Full Group Contingency — This group (n = 20) will earn vouchers based only on team (n = 4) performance. Only if all members of the team submit a negative sample (CO ≤ 4 ppm), will they each earn a voucher.
  Arms: Full Group Contingency
Behavioral: Mixed Group Contingency — This group (n = 20) will earn vouchers based on both individual and team (n = 4) performance. If an individual submits a negative sample (CO ≤ 4 ppm), s/he will earn a voucher. Additionally, bonus vouchers will be earned if all team members submit negative samples.
  Arms: Mixed Group Contingency

SUMMARY:
The purpose of the study is to develop and test an Internet-based group contingency management program designed to promote smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* self-reported smoker
* ability to use the Internet
* permission to contact applicant by phone

Exclusion Criteria:

* self-report of a history of or current severe or unstable medical or psychiatric illness that would interfere with the study
* inability to avoid high levels of ambient CO (e.g., occupational exposure; lives with a another smoker who smokes in the home)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Breath CO | 8 weeks
  Twice daily breath CO samples obtained during baseline and treatment

SECONDARY OUTCOMES:
Point prevalence measure of abstinence | at the end of treatment (approximately week 4) and at 3 month follow-up
  Abstinence will be defined as: (a) CO sample ≤ 4 ppm; (b) cotinine < 50 ng/ml; and (c) reporting not smoking, not even a puff in the last 7 days.
Duration of abstinence during treatment. | 3 weeks
  The longest duration of sustained abstinence (CO ≤ 4 ppm) based on the twice-daily breath samples during the treatment period.
Rate of social exchanges | 3 weeks
  The number of comments posted on the discussion forum during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Dallery, PhD, Principal Investigator — National Development and Research Institutes, Inc.
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - National Development and Research Institutes, New York, New York